CLINICAL TRIAL: NCT02702908
Title: Second Primary Cancers in Patients With Castration Resistant Prostate Cancer (BOCARP)
Brief Title: Second Primary Cancers in Patients With Castration Resistant Prostate Cancer
Acronym: BOCARP
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18044; EUPAS12665 (Registry Identifier: ENCEPP)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mPC: Prostate cancer patients with bone metastases (mPC)
- mCRPC: Patients with castration-resistant prostate cancer with bone metastases (mCRPC)

INTERVENTIONS:
Other:  — Historical Reference group.

SUMMARY:
This study aims at estimating the incidence of second primary malignancies as well as the overall survival among metastasized prostate cancer (mPC) and metastasized castrate-resistant prostate cancer (mCRPC) patients not treated with radium-223-dichloride.

DETAILED DESCRIPTION:
This study aims at estimating the incidence of second primary malignancies as well as the overall survival among mPC and mCRPC patients not treated with radium-223-dichloride. The source of data for this study will be the German Pharmacoepidemiological Research Database (GePaRD). A retrospective cohort study covering the time period from 2004 to 2013 will be conducted. The study population will comprise CRPC patients developing bone metastases. These patients will be followed up for the occurrence of second primary malignancies, end of study, or death due to any cause. As this study serves as a historical control group for a single-arm observational study, incidence rates of second primary malignancies obtained from these studies will be compared by the standardized incidence ratio using results from this study as a reference.

ELIGIBILITY:
Inclusion Criteria:

* Members of the mPC cohort will have to fulfill all of the following criteria:

  * Valid information on sex, age and the region of residence
  * A period of at least 12 months of continuous insurance preceding cohort entry
  * Diagnosis of PC (ICD-10 Code C61) in the study period (01-Jan-2004 to 31-Dec-2011)
  * Diagnosis of bone metastases (ICD-10 Code C79.5) in the enrolment period (01-Jan-2005 to 31-Dec-2011)
  * In addition to the criteria of the mPC cohort, members of the mCRPC will additionally have to fulfill:
  * One of the following in the enrolment period and before or at the same time with bone metastases

    * Discontinuation of the initial chemical castration, change of the agent or modality of the Androgen deprivation therapy (ADT), or start of treatment for advanced Prostate cancer (PC) after the primary ADT.
    * Surgical castration and initiation of ADT treatment
    * Treatment with medication specific to mCRPC.

Exclusion Criteria:

* Patients will be excluded from the mPC and from the mCRPC populations if they meet one of the following criteria:

  * First PC diagnosis later than 2 months after the diagnosis of bone metastases, or
  * Use of any radiopharmaceuticals for bone metastases (e.g., samarium, strontium, rhenium, radium)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of mPC patients (prostate cancer patients with bone metastases) and a subgroup of patients who can be regarded as mCRPC patients (castration-resistant prostate cancer patients with bone metastases).
Sampling Method: Non-Probability Sample
Enrollment: 6442 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Incidences of Second primary malignancies are characterized by the following ICD-10 codes: C00-C76, C81-C96, D00-D09, D37-D48. | Up to 10 years

SECONDARY OUTCOMES:
Overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany